CLINICAL TRIAL: NCT06507930
Title: The COMPASSION Study: Applying Telehealth to Innovate and Strengthen Connections for Patients With Metastatic Breast Cancer Receiving Hospice Care
Brief Title: The COMPASSION Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Claire Smith, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-142
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; Unresectable Breast Carcinoma
Keywords: Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; Unresectable Breast Cancer; Hospice Care
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Cohort (No Intervention): 25 participants will complete study procedures as follows:
  * Introduction to study and survey by brief, verbal consent via phone call.
  * At 4-6 weeks: survey completion via email or phone.
- Compassion Cohort (Experimental): 25 participants will complete study procedures as follows:
  * Introduction to study and survey by brief, verbal consent via phone call.
  * At 4-6 weeks: survey completion via email or phone.
  * 4 weekly check-ins via Zoom or phone call with study team.
  Interventions: Other: Telehealth Hospice Visits

INTERVENTIONS:
Other: Telehealth Hospice Visits — Telehealth check-in appointments with oncology care team, MD, PA, NP, or hospice nurse, via HIPAA compliant telehealth platform, Zoom, or by phone call.
  Arms: Compassion Cohort

SUMMARY:
The aim of this research study is to better understand the in-home hospice experience for participants, caregivers, hospice nurses, and oncology providers by conducting telehealth check-ins between participants and caregivers and oncology care teams.

DETAILED DESCRIPTION:
The aim of this research study is to better understand the in-home hospice experience for participants, caregivers, hospice nurses, and oncology providers by conducting telehealth check-ins between participants and caregivers and oncology care teams.

Study procedures include giving verbal consent to participate and a one-time survey delivered by email or phone call.

About 200 people, which includes 50 participants, 50 caregivers, 50 hospice nurses, and about 50 oncology providers, are expected to participate in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any gender with unresectable locally advanced or metastatic breast cancer
* Eligible for in-home hospice services and referred by DFCI clinical team to in-home hospice </= 1 week before enrollment
* Ability to conduct video or phone check-ins, even if assistance required.
* Able to provide verbal consent with a willingness to take a survey at 4-6 weeks, if medically able
* Hospice setting is within Massachusetts
* Non-English language allowed but interpreter services must be present at each meeting and will be coordinated by scheduling team
* Willingness to provide a caregiver/loved one's contact information for survey contact at 4 weeks after enrollment

Exclusion Criteria:

* Unable to provide verbal consent
* Hospice care planned outside of a home setting (note: if participants start out in a home hospice setting but later transition their hospice care to an inpatient setting, enrollment is allowed as long as they started in a home setting)
* Hospice setting outside of Massachusetts
* Individuals who are under the age of 18, as this is not a project focused on pediatric patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participant Intervention Completion | Up to 4 weeks
  Feasibility of the telehealth intervention is defined as greater than or equal to 80% of enrolled participants (18 out of 25) completing greater than or equal to 66% of the planned telehealth check-ins while the participant remains alive.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Smith, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu